CLINICAL TRIAL: NCT01791985
Title: A Single Arm Phase IIa Study (With Combination SRI) to Assess the Safety & Efficacy of AZD4547 in Combination With Either Anastrozole or Letrozole in ER+ Breast Cancer Patients Who Have Progressed on Treatment With Anastrozole or Letrozole
Brief Title: AZD4547 & Anastrozole or Letrozole (NSAIs) in ER+ Breast Cancer Patients Who Have Progressed on NSAIs (RADICAL)
Acronym: RADICAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C/23/2011; 2011-000454-32 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Results first posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; AZD4547; Safety Run-In; FGFR1; ER positive breast cancer; Single arm phase IIa study
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD4547; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): NSAI (anastrozole (1mg) or letrozole (2.5mg)), orally, once daily but together with twice daily AZD4547 (80mg).
  AZD4547 will be given on an intermittent schedule of one week on / one week off.
  Interventions: Drug: AZD4547 / anastrozole or letrozole

INTERVENTIONS:
Drug: AZD4547 / anastrozole or letrozole — Patients will continue or restart the NSAI which they have progressed* on: either anastrozole (1mg) or letrozole (2.5mg), orally, once daily but together with twice daily AZD4547 (80mg).
  AZD4547 will be given on an intermittent schedule of one week on / one week off.
  *Prior to study entry, patients must have taken anastrozole or letrozole at some stage in their treatment to date for breast cancer; and shown evidence of resistance to this therapy. The NSAI does not have to be the most recent line of treatment.

SUMMARY:
This study is looking at a new drug called AZD4547 which is being tested for the treatment of oestrogen receptor positive breast cancer. AZD4547 is a drug which specifically "blocks" proteins called fibroblast growth factor receptors (FGFR1) that are involved in the processes that help cancer cells to grow. These proteins may also be responsible for the development of resistance to hormonal therapies used to treat some breast cancers. AZD4547 is not yet approved for use in breast cancer and is therefore being used in this study as a research drug.

The investigators will also test the theory that it is not necessary for high levels of FGFR1 to be present in the body to see benefit from AZD4547. (Stage 1 only)

DETAILED DESCRIPTION:
The study will be carried out in two stages. Stage 1 is to find a suitable dose of AZD4547 which can be used together with a class of drugs called nonsteroidal aromatase inhibitors (e.g. anastrozole or letrozole) i.e. a dose which does not cause too many unacceptable side effects.

Patients with hormone sensitive (oestrogen receptor positive) breast cancer, whose current treatment with anastrozole or letrozole has recently stopped working properly will be eligible for this stage.

Stage 2 will then assess the efficacy of AZD4547, based on the change in tumour size at 12 weeks (or progression if prior to week 12), when used in combination with either anastrozole or letrozole in patients with hormone sensitive (oestrogen receptor positive) breast cancer, who have progressed on treatment with either anastrozole or letrozole in any setting.

In both stages, the study will look at how well the new treatment is tolerated.

Each patient is only allowed to take part in either stage 1 or 2.

The study will be run in 9 Hospitals across England and Scotland.

ELIGIBILITY:
Inclusion Criteria Patients must fulfil all of the following criteria.

1. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
2. Aged ≥ 25 years of age (N.B. in line with other studies with AZD4574 and due to concerns of possible effects on the immature skeleton)
3. Post menopausal women. Women will be considered postmenopausal if they have had a bilateral oophorectomy or the following specific requirements apply:

   Safety run-in:
   * Women under 50 years old would be considered post-menopausal if they have been amenorrhoeic for 24 months and have follicle-stimulating hormone (FSH) and oestradiol levels in the post-menopausal range. Patients with prior exposure to depot Luteininzing hormone releasing hormones (LHRH) analogues must be 24 months or more following the last administration
   * Women aged 50 years and older would be considered post-menopausal if they have been amenorrhoeic for 12 months and patients with prior exposure to depot LHRH analogues must be 12 months or more following the last administration
   * Women rendered amenorrhoeic by adjuvant chemotherapy, who were premenopausal or perimenopausal prior to chemotherapy, must have been amenorrhoeic for at least 24 months

   Phase IIa:
   * Women under 50 years old would be considered post-menopausal if they have been amenorrhoeic for 24 months and have follicle-stimulating hormone (FSH) and oestradiol levels in the post-menopausal range.
   * Women aged 50 years and older would be considered post-menopausal if they have been amenorrhoeic for 12 months
   * Women rendered amenorrhoeic by adjuvant chemotherapy, who were premenopausal or perimenopausal prior to chemotherapy, must have been amenorrhoeic for at least 24 months
   * Perimenopausal women rendered amenorrhoeic from exposure to depot LHRH analogues*

     * Patients must have taken LHRH analogues for at least 6 months
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
5. Histological confirmation of breast cancer with documented positive oestrogen receptor status (ER+) of primary or metastatic tumour tissue according to local laboratory parameters
6. Phase IIa: Mandatory provision of tumour biopsy for assessment of oncology biomarkers
7. Fulfils criteria for previous treatment of breast cancer*:

   Safety run-in:
   * Relapse during a single regimen of adjuvant endocrine therapy with either anastrozole or letrozole or
   * Progression during first line endocrine therapy with a non-steroidal Aromatase Inhibitor (AI) for advanced breast cancer**. Co-administration of a targeted agent with the non-steroidal AI is permitted providing all toxicities have recovered to CTCAE Grade 1 or below 1 prior regimen of chemotherapy in the advanced setting is permitted. Chemotherapy administered in the adjuvant setting is permitted

   Phase IIa:

   o Progressing or progression at some point during breast cancer treatment on endocrine therapy with a non-steroidal AI.*** Co-administration of a targeted agent with the non-steroidal AI is permitted providing all toxicities have recovered to CTCAE Grade 1 or below.
   * Prior chemotherapy in the advanced and adjuvant setting is permitted.
   * Prior treatment with exemestane with or without everolimus is permitted.

     * Human Epidermal Growth Factor Receptor 2 (HER2) positive breast cancer patients should have been offered at least one prior line of HER2 directed therapy **Advanced breast cancer: metastatic disease or locally advanced disease which is not amenable to treatment with curative intent ***anastrozole or letrozole does not have to be the most recent therapy
8. Safety run-in: At least one lesion (measurable and/or non-measurable) that can be accurately assessed by CT/MRI/plain x-ray at baseline and follow up visits Phase IIa: At least one lesion ≥ 10mm in the longest diameter at baseline (or ≥ 15mm in the short axis for nodal disease) that can be accurately measured with CT/MRI at baseline and is suitable for accurate repeated measurements. Patients with bone only metastatic cancer must have a lytic or mixed lytic-blastic lesion that can be accurately assessed by CT or MRI.
9. Safety run-in: Study entry must be preceded by a minimum of 21 days of anastrozole or letrozole treatment Phase IIa: No set duration of anastrozole or letrozole treatment prior to study entry.

Exclusion Criteria

1. Treatment with any of the following:

   1. Safety run-in: more than 1 regimen of endocrine therapy for advanced breast cancer
   2. previous exposure to any FGFR inhibitor
   3. Safety run in: more than 1 prior regimen of chemotherapy for advanced breast cancer.
   4. potent inhibitors or inducers of CYP3A4 or CYP2D6, or substrates of CYP3A4 within 2 weeks prior to first dose of study treatment (3 weeks for St John's Wort)
   5. major surgery within 4 weeks prior to first dose of study treatment
   6. radiotherapy with a wide field of radiation within 4 weeks prior to first dose of study treatment; or radiotherapy with a limited field of radiation for palliation within 2 weeks before the first dose of study treatment
2. With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE grade 1 at time of starting study
3. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
4. Any evidence of severe or uncontrolled systemic diseases or active infection
5. Any of the following cardiac criteria:

   1. Resting corrected QT interval (QTc) >470 ms
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
6. Inadequate bone marrow reserve or organ function as defined by any one of the following parameters:

   Haemoglobin < 9.0 g/dL (<90.0 g/L) Absolute neutrophil count (ANC) < 1.5 x 109 /L Platelet count < 100 x 109 /L Alanine aminotransferase > 2.5 x Upper Limit of Normal (ULN) if no demonstrable liver metastases or > 5 x ULN in the presence of liver metastases Aspartate aminotransferase > 2.5 x ULN if no demonstrable liver metastases or > 5 x ULN in the presence of liver metastases Total bilirubin > 1.5 x ULN if no demonstrable liver metastases or > 3 x ULN in the presence of liver metastases Creatinine > 1.5 times ULN or creatinine clearance <50ml/min Corrected calcium > ULN Phosphate > ULN
7. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated Investigational Medicinal Product (IMP) or previous significant bowel resection that would preclude absorption of AZD4547 or anastrozole or letrozole
8. History of hypersensitivity to anastrozole or letrozole
9. History of another malignancy within 5 yrs prior to starting study treatment, except adequately treated basal or squamous cell carcinoma of the skin, carcinoma of the cervix and the disease under study
10. Any of the following ophthalmological criteria:*

    * Current evidence or previous history of retinal pigmented epithelium detachment (RPED)
    * Previous laser treatment or intra-ocular injection for treatment of macular degeneration
    * Current evidence or previous history of soft drusen, drusenoid RPE detachment and wet macular degeneration.
    * Current evidence or previous history of retinal vein occlusion (RVO)
    * Current evidence or previous history of retinal degenerative diseases (e.g. hereditary) *Patients with uncontrolled glaucoma or intra-ocular pressure >21 mmHg at screening should be referred for ophthalmological management and the condition controlled prior to first dose of study treatment.
11. Concurrent treatment with another investigational agent or use of another investigational agent within 30 days or 5 half lives, whichever is longer, preceding the first dose of study treatment
12. Concurrent treatment with prohibited medications and wash out period for that drug will not have been completed before starting study medication

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seckl, Principal Investigator — Imperial College Healthcare NHS Trust; Nicola Cresti, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust; Richard Baird, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust; Iain MacPherson, Principal Investigator — NHS Greater Glasgow and Clyde; Amitabha Chakrabarti, Principal Investigator — Poole Hospital NHS Foundation Trust; Mojca Persic, Principal Investigator — Burton Hospitals NHS Foundation Trust; Anne Armstrong, Principal Investigator — The Christie NHS Foundation Trust; Rozenn Allerton, Principal Investigator — The Dudley Group NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Queen's Hospital, Burton-on-Trent, Burton-on-Trent, Staffs
  - Russells Hall Hospital, West C8 Admin Office, 2nd Floor, Dudley, West Midlands
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Breast Cancer Research Unit, PO Box 97, Hills Road,, Cambridge
  - Greater Glasgow Health Board, Beatson West of Scotland Cancer Centre, 1053 Great Western Road,, Glasgow
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital,1st Floor, Department of Medical Oncology, Fulham Palace Road, London
  - The Christie NHS Foundation Trust, Wilmslow Road, Withington, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Sir Bobby Robson Cancer Trials Research Centre, Freeman Hospital, High Heaton, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coombes RC, Badman PD, Lozano-Kuehne JP, Liu X, Macpherson IR, Zubairi I, Baird RD, Rosenfeld N, Garcia-Corbacho J, Cresti N, Plummer R, Armstrong A, Allerton R, Landers D, Nicholas H, McLellan L, Lim A, Mouliere F, Pardo OE, Ferguson V, Seckl MJ. Results of the phase IIa RADICAL trial of the FGFR inhibitor AZD4547 in endocrine resistant breast cancer. Nat Commun. 2022 Jun 10;13(1):3246. doi: 10.1038/s41467-022-30666-0. PMID 35688802

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD4547: Participants received NSAI (anastrozole (1mg) or letrozole (2.5mg)), orally, once daily together with twice daily AZD4547 (80mg).
  AZD4547 was given on an intermittent schedule of one week on / one week off.
Period: Overall Study
Arm/Group | AZD4547
Started | 52
Completed | 44 (Eight patients (8) discontinued study treatment prior to 12 weeks or disease disease progression)
Not Completed | 8
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- AZD4547: Participants received NSAI (anastrozole (1mg) or letrozole (2.5mg)), orally, once daily together with twice daily AZD4547 (80mg).
  AZD4547 will be given on an intermittent schedule of one week on / one week off.
Arm/Group | AZD4547
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.5 [50 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 49
  Ethnicity: Black | 2
  Ethnicity: Unknown or Not reported | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 52
Smoking [Count of Participants; unit: Participants]
  Never | 29
  Past | 18
  Current | 3
  Unknown or not reported | 2
Eastern Cooperative Oncology Group (ECOG) Status [Count of Participants; unit: Participants]
  Fully active | 33
  Restricted in physically strenuous activity | 19
Tumour Grade [Count of Participants; unit: Participants] — Tumour grade describes a tumour in terms of how abnormal the tumour cells are when compared to normal cells. It also describes how abnormal the tissues look under a microscope.
  Grade 1 - the cancer cells look very similar to normal cells and are growing slowly (low grade)
  Grade 2 - the cells don't look like normal cells and are growing more quickly than normal (intermediate grade)
  Grade 3 - the cancer cells look very abnormal and are growing quickly (high grade)
  Participants
    Grade 1 or 2 | 25
    Grade 3 or 4 | 14
    Unknown | 13
ECG [Count of Participants; unit: Participants] — A standard 12-lead ECG will be performed.
  ECGs will be recorded at the following time points:
  * Screening
  * Cycle 1 day 8: 2 hours post morning dose of study medication (AZD4547 + either anastrozole or letrozole)
  * Cycle 2 day 1 (and each subsequent cycle): any time on the day of assessment
  * At discontinuation of AZD4547 + either anastrozole or letrozole therapy
  Participants
    Normal | 33
    Abnormal | 19
Echocardiogram (ECHO) / Multiplegated acquisition (MUGA) Scan [Count of Participants; unit: Participants] — An echocardiogram and / or MUGA scan to assess left ventricular ejection fraction (LVEF) will be performed at screening, Cycle 3 day 1 (± 1 week), then every 3 months (± 1 week) and finally at AZD4547 discontinuation visit.
  Participants
    Normal | 49
    Abnormal | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Safety and tolerability of AZD4547 to be used in combination with a standard dose of anastrozole or letrozole, as assessed by Dose limiting toxicity (DLT) This is the primary outcome measure in the Safety Run-In part of the study.
Time Frame: Dose limiting toxicity (DLT) assessment window - days 1 to 28 of cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4547
Number analyzed (Participants) | 52
Participants | 10

2. Primary Outcome: Proportion of Tumour Size Change at 12 Weeks (or Progression if Prior to Week 12)
Description: This is the primary outcome measure in the Randomised Phase IIa part of the study. This is the proportion of tumour size change from baseline to week 12 (or progression if prior to week 12) based on local review of results.
Time Frame: 12 weeks
Population: Out of 52 enrolled patients, 43 patients have analyzable data. Prior to week 12, there were 8 patients who discontinued study treatment prior to progression and 1 patient who had disease progression died before tumour measurements could be taken. Therefore a total of 9 patients cannot be included in the analysis of the primary outcome.
Measure: Mean (Standard Deviation); unit: Proportion of tumour size change
Arm/Group | AZD4547
Number analyzed (Participants) | 43
Proportion of tumour size change | 0.08 (0.32)
Statistical Analysis 1: Comparison: AZD4547; Proportion of change in tumour size at 12 weeks (or progression if prior to week 12), when used in combination with either anastrozole or letrozole in ER positive breast cancer patients who have progressed on treatment with either anastrozole or letrozole in any setting; Test type: Other; Mean = 0.08, Standard Deviation 0.32

3. Secondary Outcome: Proportion of Tumour Size Change at 6, 20 and 28 Weeks
Description: Proportion of tumour size change at 6, 20 and 28 weeks to assess the efficacy of AZD4547 in combination with anastrozole or letrozole. This outcome measure is based on local review.
Time Frame: 6, 20 and 28 weeks
Population: Out of 52 enrolled patients, 48 had analyzable data at 6th week, 41 at 20th week and 40 at 28th week. At specific time points, some patients may have withdrawn or already discontinued study medication.
Measure: Mean (Standard Deviation); unit: Proportion of tumuour size change
Arm/Group | AZD4547
Number analyzed (Participants) | 48
Proportion of tumuour size change
  Proportion of tumour size change at week 6 | 0.04 (0.29)
  Proportion of tumour size change at week 20: number analyzed (Participants) | 41
  Proportion of tumour size change at week 20 | 0.09 (0.36)
  Proportion of tumour size change at week 28: number analyzed (Participants) | 40
  Proportion of tumour size change at week 28 | 0.10 (0.36)

4. Secondary Outcome: Tumour Response (RECIST Criteria) at 6, 12, 20 and 28 Weeks
Description: Tumour response (RECIST criteria) at 6, 12, 20 and 28 weeks to assess the efficacy of AZD4547 in combination with anastrozole or letrozole. This outcome measure is based on local review.
Time Frame: 6, 12, 20 and 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4547
Number analyzed (Participants) | 52
Participants
  Overall response at week 6: Complete response | 0
  Overall response at week 6: Partial response | 2
  Overall response at week 6: Stable disease | 31
  Overall response at week 6: Progressive disease | 16
  Overall response at week 6: Progressive disease before scan | 1
  Overall response at week 6: Withdrawn before scan | 2
  Overall response at week 6: Scan not done or not available | 0
  Overall response at week 12: Complete response | 0
  Overall response at week 12: Partial response | 1
  Overall response at week 12: Stable disease | 18
  Overall response at week 12: Progressive disease | 8
  Overall response at week 12: Progressive disease before scan | 17
  Overall response at week 12: Withdrawn before scan | 6
  Overall response at week 12: Scan not done or not available | 2
  Overall response at week 20: Complete response | 0
  Overall response at week 20: Partial response | 2
  Overall response at week 20: Stable disease | 13
  Overall response at week 20: Progressive disease | 3
  Overall response at week 20: Progressive disease before scan | 26
  Overall response at week 20: Withdrawn before scan | 8
  Overall response at week 20: Scan not done or not available | 0
  Overall response at week 28: Complete response | 0
  Overall response at week 28: Partial response | 2
  Overall response at week 28: Stable disease | 10
  Overall response at week 28: Progressive disease | 1
  Overall response at week 28: Progressive disease before scan | 30
  Overall response at week 28: Withdrawn before scan | 9
  Overall response at week 28: Scan not done or not available | 0

5. Secondary Outcome: Objective Response at 6, 12, 20 and 28 Weeks
Description: Objective Response at 6, 12, 20 and 28 weeks to assess the efficacy of AZD4547 in combination with anastrozole or letrozole. The Objective Response Rate (ORR) is defined as the proportion of overall complete response (CR) and overall partial response (PR) among all patients who receive at least one dose of study treatment. This outcome measure is based on local review.
Time Frame: 6, 12, 20 and 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4547
Number analyzed (Participants) | 52
Participants
  Objective response at week 6 | 0
  Objective response at week 12 | 2
  Objective response at week 20 | 3
  Objective response at week 28 | 3

6. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) was defined as the time from study enrolment to first evidence of progression. Progression is defined as overall progressive disease identified at follow-up or confirmed disease progression at the end of the trial or death.
Time Frame: 42 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD4547
Number analyzed (Participants) | 52
months | 3.1 [2.4 to 6.2]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected throughout the study, from the point that the RADICAL team confirmed patient eligibility until the end of patient follow-up, 42 months
Arm/Group | AZD4547
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 10/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4547 (N=52)
Fractured femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Fractured bone (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Unsteadiness on feet (Nervous system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Surgical or medical procedure - prolongation of hospital stay (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4547 (N=52)
Anaemia (Blood and lymphatic system disorders) | 7 (9)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2)
Metastases to lymph nodes (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7)
Bradycardia (Cardiac disorders) | 2 (2)
Cardiac aneurysm (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Corneal erosion multiple (Eye disorders) | 1 (1)
Corneal oedema (Eye disorders) | 1 (1)
Detachment of macular retinal pigment epithelium (Eye disorders) | 1 (1)
Detachment of retinal pigment epithelium (Eye disorders) | 9 (14)
Dry eye (Eye disorders) | 9 (10)
Eye disorder (Eye disorders) | 2 (2)
Eye pruritus (Eye disorders) | 1 (1)
Growth of eyelashes (Eye disorders) | 1 (1)
Increased intraocular pressure (Eye disorders) | 1 (1)
Iritis (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 2 (4)
Lacrimation increased (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Maculopathy (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (1)
Relative afferent pupillary defect (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Retinal pigment epitheliopathy (Eye disorders) | 4 (6)
Ulcerative keratitis (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 3 (3)
Visual impairment (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (7)
Constipation (Gastrointestinal disorders) | 20 (23)
Diarrhoea (Gastrointestinal disorders) | 16 (30)
Dry mouth (Gastrointestinal disorders) | 23 (30)
Dyspepsia (Gastrointestinal disorders) | 12 (17)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Glossodynia (Gastrointestinal disorders) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Hypogeusia (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 6 (14)
Nausea (Gastrointestinal disorders) | 21 (26)
Oesophagitis (Gastrointestinal disorders) | 2 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Oropharyngeal pain (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 8 (11)
Tongue coated (Gastrointestinal disorders) | 1 (1)
Tongue eruption (Gastrointestinal disorders) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 4 (6)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (10)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 12 (20)
Influenza like illness (General disorders) | 1 (1)
Lethargy (General disorders) | 7 (9)
Mucosal inflammation (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 3 (3)
Wound secretion (General disorders) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (2)
Oral candidiasis (Infections and infestations) | 5 (6)
Oral herpes (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Viral pharyngitis (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (15)
Aspartate aminotransferase increased (Investigations) | 9 (16)
Blood albumin decreased (Investigations) | 5 (13)
Blood alkaline phosphatase increased (Investigations) | 8 (12)
Blood bilirubin increased (Investigations) | 2 (4)
Blood calcium decreased (Investigations) | 1 (1)
Blood calcium increased (Investigations) | 7 (9)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2)
Blood glucose increased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 5 (5)
Blood magnesium increased (Investigations) | 1 (2)
Blood phosphorus decreased (Investigations) | 5 (7)
Blood phosphorus increased (Investigations) | 17 (30)
Blood potassium decreased (Investigations) | 1 (2)
Blood pressure increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Calcium phosphate product increased (Investigations) | 7 (11)
Carbohydrate antigen 15-3 increased (Investigations) | 1 (1)
Dermatologic examination abnormal (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (5)
Platelet count increased (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Weight decreased (Investigations) | 5 (6)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2)
White blood cells urine (Investigations) | 1 (1)
Aphagia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 10 (17)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 10 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibroma (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ageusia (Nervous system disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 15 (17)
Headache (Nervous system disorders) | 5 (5)
Hypoaesthesia oral (Nervous system disorders) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 3 (5)
Depression (Psychiatric disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 9 (15)
Breast atrophy (Reproductive system and breast disorders) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 1 (1)
Breast inflammation (Reproductive system and breast disorders) | 1 (1)
Genital discharge (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (25)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Contusion (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (9)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 4 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 8 (8)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Nail infection (Skin and subcutaneous tissue disorders) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 6 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (4)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Paronychia (Skin and subcutaneous tissue disorders) | 3 (4)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1)
Corrective lens user (Social circumstances) | 1 (1)
Breast operation (Surgical and medical procedures) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Epistaxis (Vascular disorders) | 9 (12)
Eye contusion (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No